CLINICAL TRIAL: NCT04919720
Title: RESPOND Study (Rescue for Emergency Surgery Patients Observed to uNdergo Acute Deterioration)
Brief Title: Rescue for Emergency Surgery Patients Observed to uNdergo Acute Deterioration
Acronym: RESPOND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); University of Michigan (Other); University of Southern California (Other); University of Leicester (Other); University of Birmingham (Other); Jonkoping University (Other); LP Human Factors Ltd (Unknown); Chelsea and Westminster NHS Foundation Trust (Other); HUMAN FACTORS EVERYWHERE (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESPOND NIHR200868
Record Dates: First submitted 2021-03-22; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-03

CONDITIONS: Failure to Rescue; Emergencies
Keywords: Emergency General Surgery; Safety II; Human Factors and Ergonomics; Failure to Rescue; Laparotomy
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Step-wedge, cluster-randomised trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human Factors Interventions (Other): A 'bundle' of human factors interventions designed to improve response to deteriorating patients.
  Interventions: Behavioral: FRAM Model and Human Factors/Quality Improvement Intervention

INTERVENTIONS:
Behavioral: FRAM Model and Human Factors/Quality Improvement Intervention — The group will use semi-structured interviews and ethnographic observations to inform development of a Functional Resonance Analysis Method (FRAM) model of the process for rescue of deteriorating patients in EGS, using information from 3 hospitals. A focus group approach will be used in co-designing reform of the system for responding to post-operative deterioration, working with small groups of frontline clinical staff from relevant areas in the three Trusts involved.

SUMMARY:
This is a Five Year programme designed to identify and evaluate human factors interventions to improve the response to patients deteriorating following emergency surgery.

The programme comprises four work packages:

Work Package 1: Qualitative interviews and observations to analyse current rescue systems; Work Package 2: Identify and co-design interventions to improve rescue systems,involving both staff and patients and carers; Work Package 3: Mixed-methods feasibility trial across 3 sites in England, Work Package 4: Step-wedge randomised control trial based across 24 hospital sites in England, evaluating efficacy of interventions in improving response to deteriorating patients.

DETAILED DESCRIPTION:
Patient safety researchers study problems in healthcare systems which harm patients. The investigators wish to study a healthcare situation where system problems are costing lives. In Emergency General Surgery (EGS), dealing mainly with patients with severe abdominal pain, the death rate after abdominal surgery to find out what's wrong (called 'laparotomy') is 5 times higher than for similar routine surgery. Studies of serious complications after major operations show that when patients deteriorate after surgery, their chances of survival depend on how quickly and how well clinical teams react. The investigators plan to analyse how EGS teams currently treat deteriorating patients, and help them develop and test better response systems. Up to 3000 deaths per year could be avoided if these systems were improved . Human Factors science analyses how complex work systems succeed or fail, and how to improve them. The investigators will conduct a Human Factors analysis of real life responses to deterioration in EGS laparotomy patients, examining how staff actually deal with deteriorating patients (referred to as "work as done"), and how this differs from official guidelines (referred to as "work as imagined"). A modern approach to Human Factors called "Safety II" studies both strengths and weaknesses of systems to design solutions. The investigators will use this method to analyse current EGS rescue systems, and develop a new system for managing deterioration, including ways of involving patients or carers effectively. The investigators will test and modify this system until it can be shown that it improves team performance during rescue. Once it appears stable and effective, the investigators will test it in a multi-hospital trial. Hospitals will start using the new system at different dates (decided by chance), and the investigators will compare their performance before and after they start.

The investigators will study the cost-effectiveness of the intervention and analyse what worked well and why, to make sure the lessons are learned effectively.

ELIGIBILITY:
Inclusion Criteria:

* Senior Medical staff in EGS and in other departments and disciplines with important roles in rescue (Anaesthetics, Gastroenterology, Interventional Radiology, Intensive Treatment Unit)
* Junior medical staff in EGS (First Year 1 and 2, Core trainee and Surgical Trainee 3 + grades)
* Senior nursing staff in EGS and other relevant departments (Theatres, Intensive Treatment Unit/outreach)
* Recovered patients or their carers

Exclusion Criteria:

* Patients lacking mental capacity
* Patients who cannot communicate in English AND for whom translation facilities cannot be secured
* Patients with documented PTSD (Post Traumatic Stress Disorder) related to their experience of complications after laparotomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9064 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Improvement in response to deterioration | 12 months
  Reduction in ratio of mortality to complications
Improved Effectiveness of response to deterioration | 12 months
  Number, severity and duration of Modified Early Warning Score (MEWS) system alerts,
Improved Effectiveness of response to deterioration | 12 months
  Average timings for initial response to MEWS triggers
Improved Effectiveness of response to deterioration | 12 months
  Average timings for the segments of the MEWS response process
Improved quality of response to deterioration | 12 months
  Qualitative interview data with senior surgeons showing comparison of response quality and success in cases where patient or carer alerts were present with those where they were not
Improved effectiveness of response to deterioration | 12 months
  Number of specialist interventions following emergency laparotomy

SECONDARY OUTCOMES:
Improvement in mortality of emergency laparotomy patients | 12 months
  reduction in mortality of emergency laparotomy patients
Improvement in recovery of emergency laparotomy patients | 12 months
  Reduction in ITU stay and overall hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Peter McCulloch, MBChB, MD, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Professor Peter McCulloch, Oxford, Oxfordshire
  - Buckinghamshire Healthcare NHS Trust, Stoke Mandeville

IPD SHARING:
Plan to Share IPD: No